CLINICAL TRIAL: NCT03255889
Title: Absorption and Tolerability Studies of an Emulsion Containing the Coconut Oil-derived Glycerol Tridecanoate in Healthy Men
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Expiry of grant funding
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Principal Investigator, Obstetrics & Gynaecology, Professor, National University Hospital, Singapore
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GT2016
Record Dates: First submitted 2017-08-13; First posted 2017-08-21 (Actual); Last update posted 2017-12-07 (Actual); Status verified 2017-12

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Safety; Tolerability; Pharmacokinetics; Absorption
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Active Comparator): Glyceryl Tridecanoate emulsion, single doses (5 g, 10 g, 20 g) to 3 cohorts
  Interventions: Drug: Glyceryl Tridecanoate
- Placebo (Placebo Comparator): Sunflower oil emulsion, single doses (5 g, 10 g, 20 g) to 3 cohorts
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Glyceryl Tridecanoate — Glyceryl Tridecanoate (GT) is the triglyceride form of decanoic acid (DA), a C10 fatty acid. GT belongs to the class of medium chain triglycerides (MCT), which has been accepted as a Generally Recognized As Safe food product by FDA. Decanoic acid, also known as capric acid, occurs naturally in coconut oil (8 - 10%) and palm kernel oil (4%).
  Other Names: GT
  Arms: Active
Other: Placebo — Sunflower oil emulsion of equal calories.
  Arms: Placebo

SUMMARY:
The primary aim of the study is to test safety and tolerance of oral intake of GT oil in the form of a non-diary based emulsion (10g of GT per emulsion) in healthy men. This will be a single center study, and the recruitment is expected to happen over a 1-2- month's period.

DETAILED DESCRIPTION:
Polycystic Ovarian Syndrome (PCOS) is a hormonal disorder contributing to infertility in women. PCOS is also associated with Insulin resistance (IR) occurring at a high incidence rate of 50-70%. IR is a condition in which your body loses sensitivity to insulin requiring higher levels of it to maintain normal glucose levels in blood which hormones production from ovaries. Studies have demonstrated that the prevalence of the metabolic syndrome which is a cluster of condition such as increased blood pressure, high blood sugar, excess body fat around the waist, and abnormal cholesterol in women with PCOS is significantly higher than that of the general population. Medications that improve insulin sensitivity, such as thiazolidinediones (TZDs) and Metformin, an insulin sensitizer have been used in treating women with PCOS. Metformin major side effects consist of nausea, vomiting and gastrointestinal distress. TZDs are withdrawn from the market due to their adverse effect profile, which includes liver toxicity, weight gain, swelling due to water retention and cardiovascular diseases. As current treatment options are inadequate, there is a clinical need to identify new treatment regimens with a reduced adverse effect profile to improve the management of PCOS and its related metabolic syndrome.

Glyceryl Tridecanoate (GT) is a medium chain triglyceride (MCT); a form of dietary fat, which has a long history of safe use in in foods, drugs, cosmetics, can even be provided via the veins in individuals requiring supplemental nutrition. Decanoic acid, also known as capric acid, occurs naturally in coconut oil (8 - 10%) and palm kernel oil (4%). Importantly, the published findings show that oral administration of GT, the triglyceride form of decanoic acid, can improve insulin sensitivity and storage and breakdown of fat in animal models of diabetes. Notably, in the investigators' recent findings, DA could reduce androgen production and alleviate PCOS like symptoms in a test-induced PCOS rat model. Hence, there is a high likelihood that GT can improve the management of PCOS without the undesirable side effects that are observed with the thiazolidinediones.

The primary aim of the study is to test safety and tolerance of oral intake of GT oil in the form of a non-diary based emulsion (10g of GT per emulsion) in healthy men. This will be a single center study, and the recruitment is expected to happen over a 1-2- month's period.

ELIGIBILITY:
Inclusion Criteria:

* Men
* 21 - 40 years of age
* Healthy as determined by medical, physical examination and clinical laboratory results
* Weigh at least 60 kg.
* Reliable and willing to follow study procedures.
* Able to read/ understand English
* Given written informed consent approved by NUS and the Ethical Review Board governing the site.

Exclusion Criteria:

* Known allergies to coconut oil, or related compounds,
* History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, haematological, or neurological disorders capable of significantly altering the absorption, or metabolism or elimination of drugs or of constituting a risk when taking the study medication or interfering with the interpretation of data.
* History of drug abuse
* Evidence of hepatitis B infection
* Given a blood donation of more than 450 mL in the last 3 months or any blood donation within the last month.
* Intend to use over-the counter or prescription medication known to affect reproductive or metabolic functions (e.g. hormonal pills, metformin and etc.) including steroidal preparations or intend to use vitamin, mineral, herbal or dietary supplements or intend to consume GT health supplements during the study
* Participants will be advised to avoid consuming coconut oil, or palm oil or any food products/ health supplements containing any of these oils during the study and 3 days prior to the study.

Ages: 21 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-08-28 (Estimated); Primary Completion 2017-09-24 (Estimated); Study Completion 2018-03-28 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events/severe events | 8 to 10 days
  Incidence and severity of adverse events/serious adverse events based on history, physical examination and vital signs and clinical chemistry

SECONDARY OUTCOMES:
Decanoic acid | 3 months
  Serum will be extracted from blood samples for measurement of decanoic acid using gas chromatography-mass spectrometry (GC/MS)

CONTACTS AND LOCATIONS:
Overall Officials: Eu Leong Yong, MD & PhD, Principal Investigator — National University Hospital, Singapore
Locations (1):
- Investigational Medicine Unit, National University Health System, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No